CLINICAL TRIAL: NCT01180764
Title: Effects of Lovaza Monotherapy vs. Placebo on Composition and Function of HDL and Other Lipoproteins, and on Other Lipid-Related Parameters
Brief Title: Effects of Lovaza on High Density Lipoprotein (HDL) Composition and Function in Hypertriglyceridemia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawn for administrative reasons.
Sponsor: University of Utah (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Eliot A. Brinton, MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00040562
Record Dates: First submitted 2010-05-17; First posted 2010-08-12 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2011-07

CONDITIONS: Hypertriglyceridemia
Keywords: hypertriglyceridemia; omega-3 acid ethyl esters; high-density lipoproteins; fish oil
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lovaza (Experimental): Lovaza 4g po qd
  Interventions: Drug: Lovaza (Omega-3 acid ethyl esters)
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lovaza (Omega-3 acid ethyl esters) — 1g capsules, 4 capsules po daily
  Other Names: Lovaza
  Arms: Lovaza
Drug: Placebo — Placebo matching active lovaza, 1 g capsules, 4 capsules po daily
  Arms: Placebo

SUMMARY:
Study hypothesis: Lovaza (purified prescription fish oil) is likely to help HDL (the "good cholesterol") work better.

Study summary: We are testing effects of Lovaza versus placebo, on various aspects of HDL and other lipoproteins, in patients with high triglyceride levels.

Study funding: This study is being funded by an investigator-initiated research grant from Glaxo Smith Kline.

ELIGIBILITY:
Inclusion criteria:

* Fasting TG 500-2000 mg/dL (off of TG-lowering medications-see below)
* Age 35-75 years

Exclusion criteria:

* Use of Lovaza (2g/d or more) or high-dose dietary supplement omega-3 oil (4g/d or more) in the past 2 months
* Use of lipid therapy (statin, ezetimibe, fibrate, BAS, or niacin at therapeutic dose, 1g/d or higher) in the past 3 weeks (washout of prior therapy permitted)
* Anticipated need to change type or dose of BP medicine (all types allowed), of lipid-active diabetes medication (thiazolidinedione), of oral estrogen (BCP or HRT), or glucocorticoid during the study (16 + 2 weeks = 18 weeks total)
* Excess ethanol consumption (regular intake >4 drinks/d, or binges of >8 drinks at once for men, half these levels for women)
* Poorly controlled diabetes mellitus (A1c >9%)
* History of acute or chronic pancreatitis
* Use of exenatide (Byetta) or sitagliptin (Januvia), medications believed to increase the risk of acute pancreatitis
* History of significant unexplained or uncontrolled bleeding or bruising
* Poorly controlled blood pressure (>140/90mmHg, with or without treatment)
* Poorly controlled thyroid disease (TSH outside of normal range)
* Hepatic disease (ALT > 2.5x ULN, Dx of hepatitis or cirrhosis)
* Any contraindication or prior adverse reaction to Lovaza
* Active cancer (except basal cell or squamous cell skin cancer)
* Pregnancy, plan/desire to become pregnant, breast feeding
* Inability or unwillingness to provide informed consent

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
HDL Composition | 12 weeks
  HDL composition (protein and lipid) by size (gel filtration column)

SECONDARY OUTCOMES:
HDL cholesterol composition by density subfraction | 12 weeks
  HDL composition by density gradient ultracentrifugation
Safety | 12 weeks
  Transaminases and glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Eliot A Brinton, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States